CLINICAL TRIAL: NCT03139786
Title: Prospective Follow-up of a Cohort of Patients With Aortic Valve Bicuspidia: Multicentre Study
Brief Title: Follow-up of a Cohort of Patients With Aortic Valve Bicuspidia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2012_843_0014
Record Dates: First submitted 2017-04-10; First posted 2017-05-04 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Aortic Valve, Bicuspid
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Study the natural history of bicuspid — Study the natural history of bicuspid

SUMMARY:
The aortic valve bicuspidia (BVA) is a congenital condition corresponding to the presence of 2 sigmoids instead of 3. This is the most common cardiac congenital anomaly affecting 0.5 to 2% of the population The general rule. BVA may be associated with structural damage to the ascending aorta, which exposes BVA patients to a risk of developing ascending aortic aneurysm and acute aortic accidents. Recent data from the literature have revealed that the natural history of BVA is marked by a possible development towards significant valvulopathy and / or an ascending aortic aneurysm often requiring surgical treatment. However, the natural history of bicuspid disease remains poorly understood and the prognostic factors for progression to severe valvulopathy and / or aneurysmal dilatation of the ascending aorta remain to be determined.

ELIGIBILITY:
Inclusion Criteria:

* All patients examined in the echocardiography laboratory whose objective examination was a bicuspid valve of the aortic valve
* Bicuspidia may be formerly known

Exclusion Criteria:

* Refusal to participate
* Patients who had already undergone bicuspid surgery or ascending aorta before being examined at the echocardiography laboratory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic bicuspidia examined in the echocardiography laboratory at one of the participating centers will be systematically eligible to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2011-10-14 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Analysis of 10 year mortality in cardiac surgery in a patient with bicuspid | 10 years
  Analyzing the natural history of Bicuspidia

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France